CLINICAL TRIAL: NCT01709786
Title: Non-Invasive Hemoglobin Monitoring in the Patient With Suspected Hemorrhage
Brief Title: Non-Invasive Hemoglobin Monitoring in Patients With Hemorrhage
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Betty Tsuei, Professor of Surgery, University of Cincinnati
Other Study IDs: Tsuei-2012-06
Record Dates: First submitted 2012-10-12; First posted 2012-10-18 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-05

CONDITIONS: Hemorrhage
Keywords: Hemorrhage; Hemoglobin; Non-invasive monitoring; Medical device accuracy
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Suspected Hemorrhage: There is a single group of patients in this study -- those with suspected hemorrhage who satisfy the inclusion and exclusion criteria. The same set of measurements will be take from each patients and those measurements will be compared with one another to determine accuracy.

SUMMARY:
This study will evaluate the accuracy of two rapid methods of measuring hemoglobin in patients with suspected hemorrhage. These methods will be compared with standard laboratory measurements.

DETAILED DESCRIPTION:
Anemia and bleeding are major causes of morbidity and mortality in both surgical and nonsurgical patients. The current standard of care for monitoring patients at risk for bleeding is serial measurement of hemoglobin levels. At present, the photometric cyanmethemoglobin method is the most widely used technique for monitoring hemoglobin in the lab, and is currently the gold standard. However, this method has potential for delay before final results are obtained.

Immediate hemoglobin measurements are available with portable point-of-care devices such as the iSTAT, which can produce a measurement of hemoglobin concentration in less than 1 minute. Unfortunately, the accuracy of this device has been reported to vary with hemoglobin level, and as such may not be as accurate in detecting blood loss when compared with the gold standard of laboratory analysis.

Recently, a noninvasive, spectrophotometry-based monitoring technology has been developed. This novel technology measures the differential optical density of wavelengths of light passed through the finger in a method similar to conventional pulse oximetry. While some studies have reported that this device appears to be accurate in patients undergoing elective surgical procedures, more recent work suggests that this accuracy degrades with increased blood loss, lower oximeter signal quality and lower absolute Hgb values.

We will evaluate the accuracy of point-of-care and non-invasive SpHb measurements and utility of continuous hemoglobin monitoring in an intensive care unit setting. If these methods of rapid hemoglobin measurement can be validated in patients at risk for ongoing hemorrhage, use of this technology may result in earlier detection of ongoing hemorrhage, expedite appropriate treatment, and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* admitted to surgical intensive care unit (SICU), and
* at risk of ongoing bleeding, and
* requires serial CBC measurements

Exclusion Criteria:

* < 18 years of age, or
* a prisoner, or
* unable to have pulse oximetry readings (due to injuries, burns, amputations, or related problems)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Surgical Intensive Care Unit of University Hospital, Cincinnati will be eligible for this study if they are at risk of ongoing bleeding and require serial CBC measurements. A patient will not be eligible if he or she is:(1) less than 18 years of age, (2) a prisoner, or if (3) clinicians are unable to take pulse oximetry readings due to injuries, burns, amputations, or related problems.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van KAMPEN E, ZIJLSTRA WG. Standardization of hemoglobinometry. II. The hemiglobincyanide method. Clin Chim Acta. 1961 Jul;6:538-44. doi: 10.1016/0009-8981(61)90145-0. No abstract available. PMID 14453500
- [Background] International committee for standardization in haematology. Recommendations for haemoglobinometry in human blood. Br J Haematol. 1967 Apr;13:71-5. doi: 10.1111/j.1365-2141.1967.tb00751.x. No abstract available. PMID 5608692
- [Background] Gayat E, Aulagnier J, Matthieu E, Boisson M, Fischler M. Non-invasive measurement of hemoglobin: assessment of two different point-of-care technologies. PLoS One. 2012;7(1):e30065. doi: 10.1371/journal.pone.0030065. Epub 2012 Jan 6. PMID 22238693
- [Background] May JM. Vitamin C transport and its role in the central nervous system. Subcell Biochem. 2012;56:85-103. doi: 10.1007/978-94-007-2199-9_6. PMID 22116696
- [Background] Butwick AJ, Hilton G, Riley ET, Carvalho B. Non-invasive measurement of hemoglobin during cesarean hysterectomy: a case series. Int J Obstet Anesth. 2011 Jul;20(3):240-5. doi: 10.1016/j.ijoa.2011.03.009. Epub 2011 Jun 2. PMID 21640577
- [Background] Hahn RG, Li Y, Zdolsek J. Non-invasive monitoring of blood haemoglobin for analysis of fluid volume kinetics. Acta Anaesthesiol Scand. 2010 Nov;54(10):1233-40. doi: 10.1111/j.1399-6576.2010.02321.x. PMID 21039345
- [Background] Myers D, McGraw M, George M, Mulier K, Beilman G. Tissue hemoglobin index: a non-invasive optical measure of total tissue hemoglobin. Crit Care. 2009;13 Suppl 5(Suppl 5):S2. doi: 10.1186/cc8000. Epub 2009 Nov 30. PMID 19951386
- [Background] Santora RJ, Moore FA. Monitoring trauma and intensive care unit resuscitation with tissue hemoglobin oxygen saturation. Crit Care. 2009;13 Suppl 5(Suppl 5):S10. doi: 10.1186/cc8008. Epub 2009 Nov 30. PMID 19951382
- [Background] Lamhaut L, Apriotesei R, Combes X, Lejay M, Carli P, Vivien B. Comparison of the accuracy of noninvasive hemoglobin monitoring by spectrophotometry (SpHb) and HemoCue(R) with automated laboratory hemoglobin measurement. Anesthesiology. 2011 Sep;115(3):548-54. doi: 10.1097/ALN.0b013e3182270c22. PMID 21716091
- [Background] Applegate RL 2nd, Barr SJ, Collier CE, Rook JL, Mangus DB, Allard MW. Evaluation of pulse cooximetry in patients undergoing abdominal or pelvic surgery. Anesthesiology. 2012 Jan;116(1):65-72. doi: 10.1097/ALN.0b013e31823d774f. PMID 22133758
- [Derived] Tsuei BJ, Hanseman DJ, Blakeman MJ, Blakeman TC, Yang SH, Branson RD, Gerlach TW. Accuracy of noninvasive hemoglobin monitoring in patients at risk for hemorrhage. J Trauma Acute Care Surg. 2014 Sep;77(3 Suppl 2):S134-9. doi: 10.1097/TA.0000000000000326. PMID 25159346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Suspected Hemorrhage
Started | 88
Completed | 88
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adult patients (>18 years of age) with the potential for hemorrhage and who were admitted to the Surgical Intensive Care Unit of a tertiary referral, Level I verified trauma center.
Arm/Group | Patients With Suspected Hemorrhage
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 69
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: CBC Hemoglobin Measurement Compared to Non-invasive Radical-7 Measurement
Description: Whenever blood was drawn for laboratory measurement of serum hemoglobin, we used one drop of blood to make point-of-care measurements using the CDC and Radical-7 methods.
  For purposes of reporting outcomes measures, we took an equally weighted average of measurements on each device (i.e., all measurement occasions on all patients). These are the means reported in the Outcome Measures Data Table.
Time Frame: n ≥ 1 measurements were taken each day. All measurements (n ≥ 7) from ICU Days 1-7 were used in Bland-Altman analysis, equally weighted.
Measure: Mean (95% Confidence Interval); unit: grams per deciliter
Groups:
- Radical-7 Hemoglobin: Radical-7 hemoglobin measurement
- CBC Hemoglobin: CBC hemoglobin measurement
Arm/Group | Radical-7 Hemoglobin | CBC Hemoglobin
Number analyzed (Participants) | 88 | 88
grams per deciliter | 10.7 [10.6 to 10.9] | 9.2 [9.0 to 9.3]
Statistical Analysis 1: Comparison: Radical-7 Hemoglobin vs CBC Hemoglobin; Test type: Superiority or Other; Limits of agreement — p-value is not reported since Bland-Altman is not a hypothesis testing framework; Bland-Altman Analysis = 1.49 — Limits of agreement are -2.02 to 5.00. This is not a confidence interval because Bland-Altman is not a hypothesis testing framework

2. Primary Outcome: CBC Hemoglobin Measurement Compared to Non-invasive iSTAT Measurement
Description: When blood was drawn for laboratory measurement of serum hemoglobin, one drop of blood was used to make point of care measurements using the CBC and iSTAT methods.
  For purposes of reporting outcomes measures, we took an equally weighted average of measurements on each device (i.e., all measurement occasions on all patients). These are the means reported in the Outcome Measures Data Table.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: grams per deciliter
Groups:
- iSTAT Hemoglobin: iSTAT hemoglobin measurement
Arm/Group | iSTAT Hemoglobin | CBC Hemoglobin
Number analyzed (Participants) | 88 | 88
grams per deciliter | 8.5 [8.4 to 8.7] | 9.2 [9.0 to 9.3]
Statistical Analysis 1: Comparison: iSTAT Hemoglobin vs CBC Hemoglobin; Test type: Superiority or Other; Bland-Altman Analysis — p-value not reported since Bland-Altman is not a hypothesis testing framework; Limits of agreement = -0.63 — Limits of agreement are -3.44 to 2.18. This is not a confidence interval because Bland-Altman is not a hypothesis testing framework

ADVERSE EVENTS:
Time Frame: During patient's hospital stay
Groups:
- Radical-7 vs. CBC: All patients: Difference between Radical-Y hemoglobin measurement and CBC hemoglobin measurement
Arm/Group | Radical-7 vs. CBC
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No